CLINICAL TRIAL: NCT02987426
Title: Can Brief Mindfulness-oriented Interventions Improve Psychiatric Symptoms and Shorten Psychiatric Hospitalizations? A Randomized Controlled Trial
Brief Title: Can Brief-mindfulness Interventions Improve Psychiatric Symptoms?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Dr. Karl Looper, Psychiatrist-in-Chief, Jewish General Hospital Associate Professor, Department of Psychiatry, McGill University, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16230
Record Dates: First submitted 2016-04-26; First posted 2016-12-09 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Mindfulness Intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-oriented intervention (Experimental): Patients will get a mindfulness-oriented intervention daily for 10 minutes.
  Interventions: Behavioral: Mindfulness-oriented intervention
- Treatment as Usual (No Intervention): This group will continue receiving their normal inpatient psychiatric care and receive information (paper brochures) about health promotion.

INTERVENTIONS:
Behavioral: Mindfulness-oriented intervention — The 10 minutes daily sessions every weekday, will take place at the inpatient unit in groups of 10 people. The intervention will be alternating between three forms of "moving" mindfulness-oriented interventions as detailed below:
  Seated Tai Chi: patients will slowly move their arms in soft movements coordinated with slow breaths Gentle stretching: patients will slowly stretch their bodies coordinated with the breath and with awareness of physical sensations throughout the body4 Walking meditation: patients will walk slowly in no particular direction, focusing close attention on the act of walking
  Arms: Mindfulness-oriented intervention

SUMMARY:
Mindfulness-based interventions have gained increasing popularity in recent years as effective treatment for mental illness. Mindfulness is defined as paying attention in a particular way: on purpose, in the present moment, and non-judgmentally: "Being", rather than "Doing". Such mental states can improve emotional regulation through frontal cortex inhibition of otherwise dysregulated subcortical emotion-related circuits. Formal mindfulness approaches such as mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction, have been highly effective in a broad range of psychiatric disorders.

Mindfulness-oriented interventions, are potentially useful in acute psychiatric hospitalizations, since they can be delivered as group therapies and are be both cost-effective and scalable. However, such interventions have rarely been provided to patients during psychiatric hospitalizations, where patients are treated for a variety of psychiatric diagnoses, and may have unpredictable lengths of stay. Additionally, there had been concerns that longer traditional mindfulness based interventions (e.g. 30 minute silent meditation) may exacerbate acute psychosis. However, strong evidence suggests that patients with psychotic symptoms appear to be largely unaffected by shorter interventions. Similarly, MBCT have been helpful to treat other major reasons for hospitalization such as: bipolar disorder, severe anxiety, substance use disorders, and major depressive disorder.

Few studies have examined mindfulness-oriented treatments in inpatient settings, including two small studies involving mindfulness groups on an acute psychiatric inpatient ward (n<10) . Another study (n=23) offered inpatients with a diagnosis of major depressive disorder mindfulness-based activities. All studies concluded that mindfulness-oriented approaches in inpatient settings were feasible, although these needed to be brief interventions, given the risks and lack of efficacy of longer MBI (e.g. 40-minute silent meditation) in severe mental illness.

A cross-sectional study conducted by our team (n=40) demonstrated that brief group mindfulness-oriented lasting 10 minutes were very well tolerated by 92.5% of psychiatric inpatients. The remaining 7.5% of patients left the session before 10-minutes, but had no symptomatic exacerbations or adverse effects. Moreover, the 50% of patients self- reported improvements in general well-being and mood after a single 10-minute session. Having been recently admitted to the psychiatric inpatient or having a diagnosis of acute psychosis (75% of inpatients) did not affect patients' capacity to tolerate and benefit from the intervention. In this inpatient psychiatric population, we found that mindfulness-oriented interventions that were brief and involved physical movement (e.g. seated Tai Chi) were better enjoyed compared to other interventions.

Despite the growing literature in this field, data is needed on the effectiveness and health service implications of brief group mindfulness-oriented interventions in inpatient psychiatry settings. Outcome studies conducted so far cannot be interpreted reliably due to methodological flaws, including inadequate control groups, very small sample sizes (often n<10), and lack of randomization. In Canada, the direct cost of treatment for mental illness is estimated as 42.3 billion. Much of these costs are driven by psychiatric admissions. Thus, if brief mindfulness-oriented interventions are effective at lowering psychiatric symptom severity and shortening psychiatric hospitalizations, this could lead to significant cost-savings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Admitted to the Open Unit of Jewish General Hospital Psychiatric Inpatient Unit

Exclusion Criteria:

1. Acute high risk to self and others - defined by being hospitalized in the confined (locked) unit (High Care or UTT at JGH).
2. Have been diagnosed by their psychiatrist with a diagnosis of moderate-to-severe dementia that would interfere with their ability to complete self-reported questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Brief Psychiatric Rating Scale score | 1-week follow-up

SECONDARY OUTCOMES:
Inpatient Psychiatric length of stay (days) | Within 12 months

OTHER OUTCOMES:
Insomnia with Athens scale | At admission to the psychiatry unit and at 1-week follow-up
Quality of life assessed with Euro-QOL scale | At admission to the psychiatry unit and at 1-week follow-up
Psychotropic medication and "as needed" PRN medication use | At admission to the psychiatry unit and at 1-week follow-up
Likert Scale | At 1-week follow-up
  The patient's satisfaction will be assessed with a 10 point Likerts scale

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No